CLINICAL TRIAL: NCT00578227
Title: Immunogenicity and Safety Study of GSK Biologicals' HPV Vaccine (GSK-580299) Co-administered With a Commercially Available Vaccine in Healthy Female Adolescents
Brief Title: Evaluation of Safety and Immunogenicity of Co-administering Human Papillomavirus Vaccine With Another Vaccine in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110886
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-10

CONDITIONS: Infections, Papillomavirus
Keywords: Human papillomavirus infection,; cervical cancer; HPV vaccine,
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; Papillomavirus Vaccines

ARMS (3):
- Cervarix™ & Twinrix™ Group (Experimental): Subjects received 3 doses of Human Papilloma Virus (HPV) vaccine co-administered with combined Hepatitis A & Hepatitis B (HAB) vaccine (Months 0, 1 & 6).
  Interventions: Biological: Cervarix™; Biological: Twinrix ™ Paediatric
- Cervarix™ Group (Experimental): Subjects received 3 doses of HPV vaccine (Months 0, 1 & 6).
  Interventions: Biological: Cervarix™
- Twinrix™ Group (Active Comparator): Subjects received 3 doses of HAB vaccine (Months 0, 1 & 6).
  Interventions: Biological: Twinrix ™ Paediatric

INTERVENTIONS:
Biological: Cervarix™ — Three doses of vaccine administered intramuscularly with the second and third dose given one month and six months after the first dose
  Other Names: HPV vaccine; GSK Biologicals' HPV-16/18 L1 AS04
  Arms: Cervarix™ & Twinrix™ Group; Cervarix™ Group
Biological: Twinrix ™ Paediatric — Three doses of vaccine administered intramuscularly with the second and third dose given one month and six months after the first dose
  Arms: Cervarix™ & Twinrix™ Group; Twinrix™ Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Vaccination of pre-teens and adolescents, ideally before sexual debut and thus before exposure to oncogenic HPV, is a rational strategy for prevention of cervical cancer, and so HPV vaccination could complement the existing pre-adolescent/adolescent vaccination programs. Therefore, this Phase IIIb study is designed to evaluate the safety and immunogenicity of co-administering a commercially available vaccine with GSK Biologicals' HPV-16/18 L1 AS04 (Cervarix ®) vaccine as compared to the administration of either vaccine alone. This Protocol Posting has been updated in order to comply with the FDA AA, Sept 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their legally acceptable representatives (LARs) can and will comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 9 and 15 years of age (has not attained her 16th birthday) at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment. For subjects below the legal age of consent, written informed consent must be obtained from the subject's LAR, and written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must not be pregnant.
* Subjects must be of non-childbearing potential, or if the subject is of childbearing potential, she must be abstinent or use adequate contraception for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12).
* Concurrently participating in another clinical study, at any time during the study period (up to the Month 12 telephone contact), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after each dose of vaccine(s). Administration of routine vaccines may be allowed up to 8 days before the first dose
* A subject planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding women.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of components of the investigational vaccine.
* Previous vaccination against hepatitis A or B planned administration of any hepatitis A or B vaccine other than that foreseen by the study protocol during the study period.
* History of hepatitis A or B infection.
* Known exposure to hepatitis A or B within the previous 6 weeks.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 814 (Actual)
Dates: Start 2007-12-15; Primary Completion 2008-12-01 (Actual); Study Completion 2009-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- Canada (5):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Sarnia, Ontario
- Denmark (2):
  - GSK Investigational Site, Hoersholm
  - GSK Investigational Site, Odense C
- Hungary (6):
  - GSK Investigational Site, Bordány
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Hódmezővásárhely
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szombathely
- Sweden (5):
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lycksele
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Pedersen C, Breindahl M, Aggarwal N, Berglund J, Oroszlan G, Silfverdal SA, Szuts P, O'Mahony M, David MP, Dobbelaere K, Dubin G, Descamps D. Randomized trial: immunogenicity and safety of coadministered human papillomavirus-16/18 AS04-adjuvanted vaccine and combined hepatitis A and B vaccine in girls. J Adolesc Health. 2012 Jan;50(1):38-46. doi: 10.1016/j.jadohealth.2011.10.009. PMID 22188832
- [Background] Pederson C et al. Co-administration of ASO4- adjuvanted human papillomavirus- 16/18 cervical cancer vaccine with inactivated hepatitis A ans B vaccine in girls aged 9-15 years. Abstract presented at the 6th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Beunos Aires, Argentina, 19-22 November 2009.
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110886 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although the total number of enrolled subjects for this study was 814, one subject did not receive any study vaccine and was therefore not considered as started in the 'Participant Flow' section.
Period: Overall Study
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Started | 272 | 270 | 271
Completed | 267 | 268 | 267
Not Completed | 5 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group | Total
Number analyzed (Participants) | 272 | 270 | 271 | 813
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.04) | 11.2 (2.02) | 11.2 (1.99) | 11.2 (2.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 270 | 271 | 813
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Anti-hepatitis A (Anti-HAV) Antibodies
Description: Seroconversion is defined as the appearance of anti-HAV antibodies [i.e., antibody titer greater than or equal to 15 milli-international units/milliliter (mIU/mL)] in the sera of subjects seronegative (antibody titer below 15 mIU/mL) before vaccination.
Time Frame: At Month 7
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, in subjects seronegative for anti-HAV before vaccination (i.e. with antibody titer below 15 mIU/mL).
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 240 | 0 | 242
Participants | 240 |  | 242

2. Primary Outcome: Anti-Heptatis A (HAV) Antibody Titers.
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as mIU/mL.
Time Frame: At Month 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects seronegative for anti-HAV before vaccination (i.e. with antibody titer below 15 mIU/mL).
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 240 | 0 | 242
mIU/mL | 4504.2 [3993.0 to 5080.8] |  | 5288.4 [4713.3 to 5933.7]

3. Primary Outcome: Number of Subjects Seroprotected for Anti-hepatitis B Surface Antigen (Anti-HBs) Antibodies
Description: A subject seroprotected against HBs is a subject with antibody titers greater than or equal to 10 mIU/mL.
Time Frame: At Month 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects seronegative for anti-HBs before vaccination, i.e. with anti-HBs antibody titer greater than or equal to 3.3 mIU/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 178 | 0 | 161
Participants | 175 |  | 161

4. Primary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination. Cut-off values = 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Month 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects seronegative for the corresponding HPV type before vaccination, i.e. with antibody titers below 8 EL.U/mL for anti-HPV-16 antibodies and below 7 EL.U/mL for anti-HPV-18 antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 239 | 241 | 0
Participants
  Anti-HPV-16: number analyzed (Participants) | 229 | 233 | 0
  Anti-HPV-16 | 228 | 233 |
  Anti-HPV-18 | 238 | 241 |

5. Primary Outcome: Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibody Titers
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 239 | 241 | 0
EL.U/mL
  Anti-HPV-16 GMTs: number analyzed (Participants) | 229 | 233 | 0
  Anti-HPV-16 GMTs | 22993.5 [20093.4 to 26312.0] | 26981.9 [23909.5 to 30449.1] |
  Anti-HPV-18 GMTs | 8671.2 [7651.7 to 9826.6] | 11182.7 [9924.8 to 12600.1] |

6. Secondary Outcome: Anti-HBs Antibody Titers
Description: Titers are given as Geometric Mean Titers (GMTs)expressed as mIU/mL.
Time Frame: At Month 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects seronegative for anti-HBs before vaccination, i.e. with anti-HBs antibody titers below 3.3 mIU/mL.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 178 | 0 | 161
mIU/mL | 3136.5 [2436.0 to 4038.4] |  | 5646.5 [4481.3 to 7114.6]

7. Secondary Outcome: Number of Subjects Seroconverted for Anti-HBs Antibodies
Description: Seroconversion is defined as the appearance of anti-HBs antibodies (i.e., antibody titer greater than or equal to 3.3 mIU/mL) in the sera of subjects seronegative (with antibody titers below 3.3 mIU/mL) before vaccination.
Time Frame: At month 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects seronegative for anti-HBs before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 178 | 0 | 161
Participants | 175 |  | 161

8. Secondary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies in Vaccine Recipients Aged 9 Years
Description: as for outcome 4
Time Frame: At Month 7
Population: Analysis was performed in 9-year old subjects from the ATP cohort for analysis of immunogenicity, who were seronegative for the corresponding HPV type before vaccination, i.e. with antibody titers below 8 EL.U/mL for anti-HPV-16 antibodies and below 7 EL.U/mL for anti-HPV-18 antibodies.
Measure: Count of Participants; unit: Participants
Groups:
- Twinrix™ Group: Subjects received 3 doses of combined Hepatitis A & Hepatitis B (HAB) vaccine (Months 0, 1 & 6).
- 9-Year Old Cervarix Vaccine Recipients: All 9-year subjects who received 3 doses of HPV vaccine alone or co-administered with HAB vaccine.
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group | 9-Year Old Cervarix Vaccine Recipients
Number analyzed (Participants) | 0 | 0 | 0 | 161
Participants
  Anti-HPV-16: number analyzed (Participants) | 0 | 0 | 0 | 156
  Anti-HPV-16 |  |  |  | 156
  Anti-HPV-18 |  |  |  | 161

9. Secondary Outcome: Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibody Titers in Vaccine Recipients Aged 9 Years
Description: as for outcome 5
Time Frame: At Month 7
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group | 9-Year Old Cervarix Vaccine Recipients
Number analyzed (Participants) | 0 | 0 | 0 | 161
EL.U/mL
  Anti-HPV-16 GMTs: number analyzed (Participants) | 0 | 0 | 0 | 156
  Anti-HPV-16 GMTs |  |  |  | 32170.2 [27985.5 to 36980.7]
  Anti-HPV-18 GMTs |  |  |  | 12257.1 [10644.6 to 14113.9]

10. Secondary Outcome: Number of Subjects Seroconverted for Anti-HAV Antibodies
Description: Seroconversion is defined as the appearance of anti-HAV antibodies (i.e., antibody titer greater than or equal to 15 mIU/mL) in the sera of subjects seronegative (antibody titer below 15 mIU/mL) before vaccination.
Time Frame: One month after the second dose of vaccine
Population: Analysis was performed on a subset from the ATP cohort for analysis of immunogenicity, in subjects for which a blood sample was taken at Month 2 and were seronegative for anti-HAV before vaccination, i.e. with anti-HAV antibody titers below 15 mIU/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 113 | 0 | 113
Participants | 112 |  | 112

11. Secondary Outcome: Anti-HAV Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) expressed as mIU/mL.
Time Frame: One month after the second dose of vaccine
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 113 | 0 | 113
mIU/mL | 467.0 [374.4 to 582.5] |  | 513.9 [418.7 to 630.6]

12. Secondary Outcome: Number of Subjects Seroconverted and Number of Subjects Seroprotected for Anti-HBs Antibodies
Description: Seroconversion is defined as the appearance of anti-HBs antibodies (i.e., antibody titer greater than or equal to 3.3 mIU/mL) in the sera of subjects seronegative (with antibody titers below 3.3 mIU/mL) before vaccination.
  A seroprotected subject against HBs is a subject with antibody titers greater than or equal to 10 mIU/mL.
Time Frame: One month after the second dose of vaccine
Population: Analysis was performed on a subset from the ATP cohort for analysis of immunogenicity, in subjects for which a blood sample was taken at Month 2 and were seronegative for anti-HBs with antibody titers below 3.3 mIU/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 70 | 0 | 58
Participants
  Seroconverted | 68 |  | 56
  Seroprotected | 60 |  | 53

13. Secondary Outcome: Anti-HBs Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) expressed as mIU/mL.
Time Frame: One month after the second dose of vaccine
Population: Analysis was performed on a subset from the ATP cohort for analysis of immunogenicity, in subjects for which a blood sample was taken at Month 2 and were seronegative for anti-HBs before vaccination, i.e. with antibody titers below 3.3 mIU/mL.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 70 | 0 | 58
mIU/mL | 33.7 [24.9 to 45.8] |  | 43.0 [30.1 to 61.3]

14. Secondary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination. Cut-off values assessed include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: One month after the second dose of vaccine
Population: Analysis was performed on a subset from the ATP cohort for analysis of immunogenicity, in subjects for which a blood sample was taken at Month 2 and were seronegative for the corresponding HPV type before vaccination, i.e. with antibody titers below 8 EL.U/mL for anti-HPV-16 antibodies and below 7 EL.U/mL for anti-HPV-18 antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 112 | 112 | 0
Participants
  Anti-HPV-16: number analyzed (Participants) | 105 | 107 | 0
  Anti-HPV-16 | 105 | 106 |
  Anti-HPV-18 | 112 | 111 |

15. Secondary Outcome: Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibody Titers
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as EL.U/mL.
Time Frame: One month after the second dose of vaccine
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 112 | 112 | 0
EL.U/mL
  Anti-HPV-16 GMTs: number analyzed (Participants) | 105 | 107 | 0
  Anti-HPV-16 GMTs | 5215.2 [4598.2 to 5915.0] | 4967.2 [4142.5 to 5956.1] |
  Anti-HPV-18 GMTs | 4496.8 [3899.4 to 5185.8] | 4266.5 [3562.9 to 5109.0] |

16. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include injection site pain, redness and swelling. Data are presented across doses.
Time Frame: During the 7-day period (Day 0-6) following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 269 | 270 | 271
Participants
  Pain | 251 | 250 | 202
  Redness | 155 | 170 | 74
  Swelling | 146 | 137 | 56

17. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, rash, temperature [axillary route, greater than or equal to 37.5 degree Celsius (°C)] and urticaria.
Time Frame: During the 7-day period following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 269 | 270 | 271
Participants
  Arthralgia | 50 | 45 | 40
  Fatigue | 122 | 133 | 119
  Fever | 24 | 28 | 14
  Gastrointestinal | 70 | 65 | 72
  Headache | 125 | 124 | 110
  Myalgia | 103 | 99 | 75
  Rash | 18 | 21 | 12
  Urticaria | 6 | 11 | 9

18. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Throughout the active phase of the study (up to Month 7)
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 272 | 270 | 271
Participants | 22 | 23 | 31

19. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: as for outcome 18
Time Frame: Throughout the safety follow-up (from Month 7 up to Month 12)
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 272 | 270 | 271
Participants | 2 | 2 | 1

20. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse events include any adverse event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30-day period following any vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 272 | 270 | 271
Participants | 83 | 96 | 83

21. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study (up to Month 12)
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Number analyzed (Participants) | 272 | 270 | 271
Participants | 2 | 4 | 4

ADVERSE EVENTS:
Time Frame: From Day 0 up to Month 12
Arm/Group | Cervarix™ & Twinrix™ Group | Cervarix™ Group | Twinrix™ Group
Serious Adverse Events (participants affected / at risk) | 2/272 | 4/270 | 4/271
Other Adverse Events (participants affected / at risk) | 258/272 | 256/270 | 224/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix™ & Twinrix™ Group (N=272) | Cervarix™ Group (N=270) | Twinrix™ Group (N=271)
Anal abscess (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix™ & Twinrix™ Group (N=272) | Cervarix™ Group (N=270) | Twinrix™ Group (N=271)
Pain at injection site (General disorders) | 251 | 250 | 202
Redness at injection site (General disorders) | 155 | 170 | 74
Swelling at injection site (General disorders) | 146 | 137 | 56
Arthralgia (General disorders) | 50 | 45 | 40
Fever (General disorders) | 24 | 28 | 14
Gastrointestinal symptoms (General disorders) | 70 | 65 | 72
Headache (General disorders) | 125 | 124 | 110
Myalgia (General disorders) | 103 | 99 | 75
Rash (General disorders) | 18 | 21 | 12
Nasopharyngitis (Infections and infestations) | 6 | 21 | 13
Fatigue (General disorders) | 122 | 133 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.